CLINICAL TRIAL: NCT04432415
Title: Comparison of the Efficacy of Silver Diamine Fluoride Solution and Sodium Fluoride Varnish for the Prevention and Arrest of Root Caries in a Group of Older Adults
Brief Title: Comparison of Silver Diamine Fluoride and Sodium Fluoride Varnish to Prevent and Arrest Root Caries in Older Adults
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Coronavirus Pandemic
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Collaborators: Sistema para el Desarrollo Integral de la Familia (Unknown)
Responsible Party: Principal Investigator, Aida Borges, Principal investigator, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UNAMexico CIE/0810/03/2017
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Root Caries
Keywords: root caries; Fluorides; aged; incidence; Mexico; Long-Term Care
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Intervention Model Description: Participants will be assigned randomly into treatment and control group using a randomization protocol.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know which type of fluoride they are getting. Outcome assesor will not know the type of fluoride or placebo assigned to each group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Silver Diamine Fluoride (Experimental): Participants receive Annual applications of 38% SDF solution and semestral applications of artificial saliva and a personalized dental health education program.
  Interventions: Device: Silver Diamine Fluoride
- Group Sodium Fluoride Varnish (Experimental): Participants receive semestral applications of Sodium Varnish Fluoride and a personalized dental health education program.
  Interventions: Device: Soduim Fluoride Varnish
- Placebo (Placebo Comparator): Participants receive semestral apllications of artificial saliva and a personalized dental health education program.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Silver Diamine Fluoride — Annual application od Silver Diamine Fluoride
  Arms: Group Silver Diamine Fluoride
Device: Soduim Fluoride Varnish — biannual apllication of Sodium Fluoride Varnish
  Arms: Group Sodium Fluoride Varnish
Device: Placebo — biannual application of artificial saliva
  Arms: Placebo

SUMMARY:
Dental caries (coronal and root) is highly prevalent in older adults. It is important to identify and implement the most effective methods that prevent the formation of root caries lesions and inhibit existing lesions at the community level.

A clinical trial will be conducted in three groups of adults 60 years old and older, comparing the application of silver diamine fluoride solution and sodium fluoride varnish in dental root surfaces with caries and sound root surfaces. The objectives are to determine over a 30-month period which of the two agents is most effective in reducing the incidence of root caries, and which is most effective in arresting active root caries lesions.

Hypothesis: the incidence of root caries will be lower in the group of subjects treated with silver diamine fluoride compared to sodium fluoride varnish. The arrest of active root lesions will be higher when using silver diamine fluoride compared to sodium fluoride varnish.

Signed informed consent will be requested from persons 60 years and over, residents of four long-term care centers and attendees of a day care center in four central states of Mexico: Mexico City, Cuernavaca City, Oaxaca City and Toluca City. All facilities are administered by the National System for Integral Family Development (IFD), a public welfare institution that works at the federal and state levels.

Three groups will be formed (60 participants in each), two groups will be administered each of the agents, the third group will be the control group. All groups will receive dental health education (oral hygiene, instructions for care and hygiene of removable dental prosthesis, information on prevention of coronal and root caries and periodontal diseases). The preventive agents will be administered according to the manufacturer's instructions. Clinical evaluations will be carried out at baseline 6, 12, 18, 24 and 30 months. The incidence of root caries among the groups will be compared with the percentage of active root lesions that were arrested and that remained inactive.

If the greater efficacy of silver diamine fluoride is proven, it can be proposed for use in caries preventive programs for older persons, reducing the risk of tooth loss and improving quality of life. It will also serve as a guide for dental surgeon in-office decision-making regarding the method to use to prevent and limit root caries lesions in older adults at risk.

DETAILED DESCRIPTION:
There is an increase in the incidence and prevalence of chronic diseases, including oral problems in older persons. Coronal and root caries, and periodontitis represent the main causes of tooth loss, and in older adults they have a great impact on quality of life, nutritional status, social life, and the increased risk of systemic problems related to dental infectious processes. At present, older adults have more remaining teeth and dental caries is highly prevalent. It is important to investigate and implement methods that prevent the formation of new carious lesions and that arrest existing lesions. The utilization of silver diamine fluoride as a method to prevent coronal caries has been recognized and has proven to be highly effective in treating dentin hypersensitivity and arresting active lesions, also it is easy to apply. Therefore, it is important and necessary to implement methods that avoid the formation of lesions and that inhibit the root caries lesions already present.

If greater effectiveness of silver diamine fluoride in preventing and arresting active root caries is confirmed, its use in conjunction with oral health education can be proposed as a preventive method to be included in oral health programs in institutionalized persons in whom dental care and attention are less frequent. Its ease of application, the longer time between applications and its cost can facilitate better oral care. On the other hand, the results can guide professionals in clinical practice in making decisions regarding the most appropriate method to prevent and arrest root caries lesions in their patients.

Hypothesis The incidence of root caries (new root caries lesions) after 30 months will be lower on root surfaces that have been treated with silver diamine fluoride solution (38% concentration [44800 ppm]) compared to those treated with sodium fluoride varnish (5% concentration [22,600 ppm]) and to those in the control group (artificial saliva).

The number of active root caries lesions arrested at baseline will be higher in people who have been treated with silver diamine fluoride solution (38% concentration [44,800 ppm]) compared to those treated with sodium fluoride varnish (5% concentration [22600 ppm]) and with the control group (artificial saliva).

General objective:

To identify whether the annual application of silver diamine fluoride solution combined with an individualized oral health education program is more effective than biannual application of sodium fluoride varnish combined with an individualized oral health education program and a group control (artificial saliva and oral health individualized educational program) in the reduction of the incidence of root caries and in the arrest of active root caries lesions over a period of 30 months in a population of adults over 60 years of age in residents of 4 gerontological centers and a DIF day care center, in 2017-2020.

Specific objectives:

* To compare the incidence of root caries after 30 months in three groups receiving the annual application of silver diamine fluoride solution (44800 ppm), the biannual application of sodium fluoride varnish (22600 ppm) and the biannual application of artificial saliva respectively, controlling for age, gender, frequency of toothbrushing, use of dental floss, use of removable prostheses.
* To compare the number of active root carious lesions arrested at baseline after annual application of silver diamine fluoride solution (44,800 ppm) and biannual application of sodium fluoride varnish (22,600 ppm) and biannual application of artificial saliva, all combined with an individualized oral health education program, controlling by age, gender, frequency of toothbrushing, use of dental floss, use of removable prostheses.
* To design and implement an individualized oral health education program on prevention and treatment of root and coronal caries, promotion and reinforcement of toothbrushing, and the proper care and cleaning of removable prostheses.

METHODS Area: clinical research Study type: Intervention Study design: randomized controlled clinical trial. Study characteristics: prospective, longitudinal, comparative. Participant allocation: randomized Study classification: efficacy study Intervention model: parallel groups Masking: blind (participant) Main purpose: Prevention Study population Residents of four gerontological centers "Arturo Mundet" (Mexico City), "Vicente García Torres" (Mexico City), "Los Tamayo" (Oaxaca, Oaxaca) and "Olga Tamayo" (Cuernavaca, Morelos ) and a day care center in Santa Ana Tlapaltitlán (Toluca, State of Mexico). All centers are administered by the National System for Integral Family Development, a public welfare institution that works at the federal and state levels.

Sample size Three groups of size 60 are required, in a no probabilistic convenience sampling.

The administration will be carried out in the same way in the three groups using a mini applicator brush.

Control group: biannual application of artificial saliva on exposed root surfaces. Sodium Fluoride varnish: biannual application of sodium fluoride varnish (22,600 ppm) on exposed healthy root surfaces and application at baseline and biannually on active root lesions. Silver Diamine Fluoride: annual application of silver diamine fluoride solution (44800ppm) on exposed healthy root surfaces and alternate annual application of artificial saliva, as well as initial and annual application on active root lesions.

Before data collection persons will be invited to participate, the purpose of the study will be explained, and if they accept will be examined to identify whether they meet the selection criteria.

Once the participants have been selected and signed the informed consent, they will be randomly assigned to one of the three groups. The baseline questionnaire on knowledge, attitudes and practices, the clinical evaluation and the initial application of the preventive agents or placebo, and the first personalized oral health education session will be carried out.The clinical examination will be carried out in each center using a portable dental unit and artificial light.

The evaluations will be repeated at 6, 12, 18, 24 and 30 months. The examiner will be standardized for the evaluation of root caries using the International Caries Detection and Assessment System (ICDAS) for root caries, and in the assessment of dental plaque and dental calculus.

ELIGIBILITY:
Inclusion criteria:

* Adults 60 years of age and older
* At least 5 teeth with gingival recession and exposed root surfaces not indicated for extraction
* No problems performing activities of daily living
* Agree to participate and sign the informed consent.

Exclusion criteria:

* Health problems that prevent oral hygiene
* Cognitive problems that prevent understanding oral hygiene instructions
* Salivary gland diseases (hyposalivation)
* Having received radiation therapy to the head and neck
* Deafness
* Active infections of the oral mucosa
* Allergy to silver
* Stomatitis
* Allergy to colophony (component of varnishes)

Elimination criteria:

-Adults who do not return to subsequent applications of silver diamine fluoride, sodium fluoride varnish, or artificial saliva.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of root caries lesions | 30 months
  Number of new caries lesions

SECONDARY OUTCOMES:
Arrested root caries lesions | 30 months
  number of active root caries lesions arrested (non active)

CONTACTS AND LOCATIONS:
Overall Officials: Aida Borges-Yañez, PhD, Principal Investigator — Universidad Nacional Autonoma de Mexico
Locations (1):
- Centro Gerontológico Arturo Mundet, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deutsch A. An alternate technique of care using silver fluoride followed by stannous fluoride in the management of root caries in aged care. Spec Care Dentist. 2016 Mar-Apr;36(2):85-92. doi: 10.1111/scd.12153. Epub 2015 Dec 21. PMID 26687774
- [Background] Tan HP, Lo EC, Dyson JE, Luo Y, Corbet EF. A randomized trial on root caries prevention in elders. J Dent Res. 2010 Oct;89(10):1086-90. doi: 10.1177/0022034510375825. Epub 2010 Jul 29. PMID 20671206
- [Background] Zhang W, McGrath C, Lo EC, Li JY. Silver diamine fluoride and education to prevent and arrest root caries among community-dwelling elders. Caries Res. 2013;47(4):284-90. doi: 10.1159/000346620. Epub 2013 Feb 5. PMID 23392087
- [Background] Sequeira-Byron P, Lussi A. Prevention of root caries. Evid Based Dent. 2011;12(3):70-1. doi: 10.1038/sj.ebd.6400805. PMID 21979764
- [Background] Richards D. Fluoride has a beneficial effect on root caries. Evid Based Dent. 2009;10(1):12. doi: 10.1038/sj.ebd.6400627. PMID 19322220
- [Background] Twetman S, Keller MK. Fluoride Rinses, Gels and Foams: An Update of Controlled Clinical Trials. Caries Res. 2016;50 Suppl 1:38-44. doi: 10.1159/000439180. Epub 2016 Apr 22. PMID 27101002